CLINICAL TRIAL: NCT05987111
Title: Comparison of Efficacy of Two Different Pilates Exercise Methods in Individuals With Ankylosing Spondylitis: A Randomized Controlled Study
Brief Title: Pilates in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, principal investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exercise
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mat Pilates (Active Comparator): Mat Pilates Exercises
  Interventions: Behavioral: Pilates
- Reformer Pilates (Experimental): Reformer Pilates Exercises
  Interventions: Behavioral: Pilates

INTERVENTIONS:
Behavioral: Pilates — Pilates exercises were applied twice a week for 4 weeks in both groups. The sessions were supervised by an Australian Physiotherapy and Pilates Institute (APPI) certified physiotherapist as 5 minutes of warm-up, 45 minutes of exercise and 5 minutes of cool-down periods.

SUMMARY:
This study was planned to examine and compare the effectiveness of two different pilates exercise methods (mat pilates vs reformer pilates) in individuals with Ankylosing Spondylitis(AS).

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 20-65, using stable medication for at least 3 months, being sedentary (Not regularly participating in exercise activities for the past 3 months).

Exclusion Criteria:

* the presence of cardiovascular, pulmonary, orthopedic and neurological problems, another rheumatic disease, being pregnant, inability to participate in at least 75% of the exercises.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index | 10 minutes
  This index consists of 5 measurements: cervical rotation, tragus to wall distance, lumbar side flexion, modified Schober's, intermalleolar distance.
Bath Ankylosing Spondylitis Disease Activity Index | 5minutes
  BASDAI consists of 6 questions evaluating the patient's level of weakness/fatigue, spinal pain, joint pain/swelling and sensitivity to touch, and duration of morning stiffness in the last week.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 5 minutes
  This scale, which evaluates the functional limitation of AS patients in activities of daily living, consists of 10 questions.
Ankylosing Spondylitis Quality of Life Questionnaire | 5 minutes
  This questionnaire, which evaluates disease-specific quality of life, consists of 18 questions
Maastrich Ankylosing Spondylitis Enthesitis Score | 5minutes
  Its validity and reliability were defined to evaluate enthesopathy and peripheral joint involvement.
Multidimensional Assessment of Fatigue Scale | 5 minutes
  MAF scale evaluates the level of fatigue during daily activities in the last week.
Biopsychosocial Questionnaire (BETY-BQ) | 10minutes
  The BETY-BQ evaluates the biopsychosocial status of patients with rheumatic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No